CLINICAL TRIAL: NCT01465503
Title: Bivalirudin in Patient at High Risk of Bleeding Undergoing Percutaneous Coronary Interventions.
Brief Title: Novel Approaches in Preventing and Limiting Events III Trial (NAPLES III): Bivalirudin in High-risk Bleeding Patients
Acronym: NAPLESIII
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Clinica Mediterranea (Other)
Responsible Party: Principal Investigator, Carlo Briguori, MD, PhD, Chief of Interventional Cardiology, Clinica Mediterranea
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NCTCM02
Record Dates: First submitted 2011-11-01; First posted 2011-11-04 (Estimated); Last update posted 2014-04-08 (Estimated); Status verified 2014-04

CONDITIONS: Bleeding
Keywords: bleeding; percutaneous coronary intervention; heparin; bivalirudin
MeSH Terms: conditions — Hemorrhage | interventions — bivalirudin; Heparin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Unfractionated Heparin (Placebo Comparator): Patients randomized to the Control group will receive unfractionated heparin (UFH) before and during the procedure. UFH bolus will be of 70 UI/kg. If the activated clotting time measured 5 minutes after the study drug administration is lower than 270 seconds, an additional bolus of the randomised drug (UFH 20 U/kg) will be given.
  Interventions: Drug: Unfractionated Heparin
- Bivalirudin (Active Comparator): Patients randomized to Bivalirudin group will be treated by bivalirudin before and during the procedure. Bivalirudin will be given as bolus of 0.75 mg/kg prior to the start of the intervention, followed by infusion of 1.75 mg/kg per hour for the duration of the procedure.The infusion will be lowered to 1.0 mg/kg per hour in patients with eGFR <30 ml/min/1.73 m2.
  Interventions: Drug: Bivalirudin

INTERVENTIONS:
Drug: Bivalirudin — Patients randomized to Bivalirudin group will be treated by bivalirudin before and during the procedure. Bivalirudin will be given as bolus of 0.75 mg/kg prior to the start of the intervention, followed by infusion of 1.75 mg/kg per hour for the duration of the procedure.The infusion will be lowered to 1.0 mg/kg per hour in patients with eGFR <30 ml/min/1.73 m2.
  Other Names: Bivalirudin (Angiox; The Medicine Company - NJ 07054 U.S.A)
  Arms: Bivalirudin
Drug: Unfractionated Heparin — Patients randomized to the Control group will receive unfractionated heparn (UFH) before and during the procedure. UFH bolus will be of 70 UI/kg. If the activated clotting time measured 5 minutes after the study drug administration is lower than 270 seconds, an additional bolus of the randomised drug (UFH 20 U/kg) will be given.
  Arms: Unfractionated Heparin

SUMMARY:
Bleeding occurring during percutaneous coronary interventions (PCI has now emerged as one of the most common complication of PCI and adversely affect in-hospital, short- and long-term outcome.As bivalirudin proved its effectiveness in decreasing haemorrhagic events during PCI, its administration may be advocated in subjects deemed at high risk of bleeding.Objective of the present trial is to compare the safety and effectiveness of procedural use of bivalirudin in comparison to unfractionated heparin (UFH) in patients undergoing PCI deemed at high risk of procedural bleeding.

DETAILED DESCRIPTION:
Antithrombotic and antiplatelet therapies have been the focus of extensive clinical investigations over the past 2 decades. In PCI settings all therapies inhibiting coagulation and primary hemostasis may limit ischaemic event rates, but are associated with an increased risk of bleeding. Retrospective and registry data indicates that haemorrhage is associated with mortality in patients undergoing PCI, emphasizing the potential importance of minimizing bleeding, as well as ischemic events, bleeding has now emerged as one of the most common complication of PCI. Major bleeding and blood transfusion have been strongly associated with increased rates of in-hospital and late mortality, MI and repeat revascularization after PCI. Also minor bleeding, although represent a complication significantly less dangerous than major haemorrhages, are associated with prolonged hospitalization, increased cost and adversely affect short- and long-term outcome.

UFH is the most commonly used anticoagulant drug during PCI. Bleeding events during PCI may be in part due to the use of this drug. Bivalirudin (The Medicine's Co., Parsippany, NJ) is a synthetic direct thrombin inhibitor approved for patients with stable and unstable coronary syndromes undergoing PCI. Favourable properties of bivalirudin may minimize bleeding.

Several clinical and procedural factors have been evaluated to identify patients exposed to a higher risk of hemorrhages. Nikolsky et al. have developed a risk score (validated on REPLACE-1 and REPLACE-2 data) based on clinical variable useful to predict the incidence of major peri-procedural bleeding after contemporary PCI using the femoral approach. The clinical variables considered into this algorithm are age >55 years (integer score 4 for every 10 years over 55), female gender (integer score 3), eGFR <60 ml/min/1.73 m2 (integer score 2), pre-existing anaemia (integer score 2), and administration of low-molecular weight heparin within 48 hours (integer score 2). Global risk score 0-1 anticipated a major bleeding rate of 1.3%; a risk score 2-6 was associated with a 1.8% risk of major bleeding; a risk score 7-9 associated with a 2.7% risk if major bleeding, whereas a risk score >=10 was associated with a 5% rate of major bleeding.

Our hypothesis is that bivalirudin, compared with UFH, may provide significant benefits in term of bleeding in the selected population of patients deemed at high risk of bleeding. Our aim is thus to prove, in a double-centres, randomized, blind controlled trial enrolling patients undergoing PCI via the femoral approach, the efficacy in term of haemorrhagic events and, secondarily, the effectiveness and safety of bivalirudin by means of the study drug vs UFH.

Sample size estimation: in this high risk population we expect a rate of major and minor bleeding of >5% for the UFH group vs a 3% event rate in the bivalirudin group. Aiming for a 0.05 alpha and 0.80 power, a total of 662 patients will need to be enrolled (331 patients per group). This will be increased by about 25% (leading to a total of 830 patients) because of considerable uncertainty about expected end-point rates.

ELIGIBILITY:
Inclusion Criteria:

* • Male or female able to understand and sign a witnessed informed consent

  * Age ≥ 18 ys
  * Patients with stable (CCS 1-4) or unstable angina pectoris (but with the most recent anginal episode occurring >48 hours before the procedure) or documented silent ischemia
  * Stable Hemodynamic conditions (systolic BP > 100 HR > 40 < 100).
  * No clinical and ECG changes suggestive of ongoing acute or recent (<48 hours) myocardial infarction.
  * Bleeding risk score ≥ 10
  * Procedure planned via femoral approach
  * Double antiplatelet therapy.

4.2.2 Angiographic inclusion criteria

• Angiographic evidence of a de novo lesion > 50% requiring intervention

Exclusion Criteria:

* • Female sex with childbearing potential

  * Age <18 years
  * Ongoing or recent episode (<48 hours) of unstable coronary artery disease (including both ST-elevation and non-ST-elevation acute coronary syndromes)
  * Chronic kidney disease (estimated glomerular filtration rate <30mL/min/1.73 m2).
  * Ongoing serious bleeding or bleeding diathesis
  * Previous stroke in the last 6 months
  * Platelet count ≤100,00 per mm3
  * History of heparin- induced-thrombocytopenia
  * Known hypersensitivity or contraindication to aspirin, heparin, clopidogrel, or sensitivity to contrast which cannot be adequately pre-medicated.
  * Hemodynamic instability (systolic blood pressure < 100 mm Hg; heart rate < 40 bpm or >100 bpm; complex ventricular arrhythmias; AV block) requiring balloon counterpulsation or inotropic support.
  * The patient is simultaneously participating in another device or drug study. Patient must have completed the follow-up phase of any previous study at least 30 days prior to enrolment in this study.
  * Positive clinical history for intracranial neoplasia, AV malformation, aneurysm.
  * INR ≥ 2.0 or prothrombin time 1.2 times upper limit of normality

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 837 (Actual)
Dates: Start 2008-01; Primary Completion 2012-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
The primary end point will be the rate of in-hospital major bleeding, defined according to the REPLACE-2 criteria. | Within 24 hours
  Major bleeding are defined as intracranial, intraocular, or retroperitoneal haemorrhage, clinically overt blood loss resulting in a decrease in haemoglobin of more than 3 g/dL, any decrease in haemoglobin of more than 4 g/dL, or transfusion of 2 or more units of packed red blood cells or whole blood.

SECONDARY OUTCOMES:
Cardiac death within 30, 180 and 360 days. | At 12 months from the PCI
  Cardiac death: all deaths unless an unequivocal non-cardiac cause can be established.
New myocardial infarction | at 12 months
  1. Q wave MI will = development of a new abnormal or worsened Q-waves not present on the patient's baseline ECG.
  2. Non-Q-wave MI = as MB iso-enzyme of creatinine kinase (CK-MB)>3X ULN .
Major and minor bleeding rate | at 30 days
  1. Major bleeding = see above.
  2. Minor bleeding = clinically overt bleeding that did not meet criteria for major.
target vessel revascularization (TVR) | at 12 monhts
  TVR = revascularization procedure (repeat angioplasty or coronary bypass surgery) targeting the target vessel

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - IRCCS Policlinico Multimedica, Milan, Milan
  - Clinica Mediterranea, Naples, Naples

REFERENCES:
- [Background] King SB 3rd, Smith SC Jr, Hirshfeld JW Jr, Jacobs AK, Morrison DA, Williams DO, Feldman TE, Kern MJ, O'Neill WW, Schaff HV, Whitlow PL; ACC/AHA/SCAI; Adams CD, Anderson JL, Buller CE, Creager MA, Ettinger SM, Halperin JL, Hunt SA, Krumholz HM, Kushner FG, Lytle BW, Nishimura R, Page RL, Riegel B, Tarkington LG, Yancy CW. 2007 focused update of the ACC/AHA/SCAI 2005 guideline update for percutaneous coronary intervention: a report of the American College of Cardiology/American Heart Association Task Force on Practice guidelines. J Am Coll Cardiol. 2008 Jan 15;51(2):172-209. doi: 10.1016/j.jacc.2007.10.002. No abstract available. PMID 18191745
- [Background] Topol EJ, Mark DB, Lincoff AM, Cohen E, Burton J, Kleiman N, Talley D, Sapp S, Booth J, Cabot CF, Anderson KM, Califf RM. Outcomes at 1 year and economic implications of platelet glycoprotein IIb/IIIa blockade in patients undergoing coronary stenting: results from a multicentre randomised trial. EPISTENT Investigators. Evaluation of Platelet IIb/IIIa Inhibitor for Stenting. Lancet. 1999 Dec 11;354(9195):2019-24. doi: 10.1016/s0140-6736(99)10018-7. PMID 10636365
- [Background] Medina HM, Bhatt DL. Evolution of anticoagulant and antiplatelet therapy: benefits and risks of contemporary pharmacologic agents and their implications for myonecrosis and bleeding in percutaneous coronary intervention. Clin Cardiol. 2007 Oct;30(10 Suppl 2):II4-15. doi: 10.1002/clc.20237. PMID 18228647
- [Background] Ndrepepa G, Berger PB, Mehilli J, Seyfarth M, Neumann FJ, Schomig A, Kastrati A. Periprocedural bleeding and 1-year outcome after percutaneous coronary interventions: appropriateness of including bleeding as a component of a quadruple end point. J Am Coll Cardiol. 2008 Feb 19;51(7):690-7. doi: 10.1016/j.jacc.2007.10.040. PMID 18279731
- [Background] Moscucci M, Fox KA, Cannon CP, Klein W, Lopez-Sendon J, Montalescot G, White K, Goldberg RJ. Predictors of major bleeding in acute coronary syndromes: the Global Registry of Acute Coronary Events (GRACE). Eur Heart J. 2003 Oct;24(20):1815-23. doi: 10.1016/s0195-668x(03)00485-8. PMID 14563340
- [Background] Feit F, Voeltz MD, Attubato MJ, Lincoff AM, Chew DP, Bittl JA, Topol EJ, Manoukian SV. Predictors and impact of major hemorrhage on mortality following percutaneous coronary intervention from the REPLACE-2 Trial. Am J Cardiol. 2007 Nov 1;100(9):1364-9. doi: 10.1016/j.amjcard.2007.06.026. Epub 2007 Aug 16. PMID 17950791
- [Background] Anand SX, Kim MC, Kamran M, Sharma SK, Kini AS, Fareed J, Hoppensteadt DA, Carbon F, Cavusoglu E, Varon D, Viles-Gonzalez JF, Badimon JJ, Marmur JD. Comparison of platelet function and morphology in patients undergoing percutaneous coronary intervention receiving bivalirudin versus unfractionated heparin versus clopidogrel pretreatment and bivalirudin. Am J Cardiol. 2007 Aug 1;100(3):417-24. doi: 10.1016/j.amjcard.2007.02.106. Epub 2007 Jun 13. PMID 17659921
- [Background] Stone GW, Witzenbichler B, Guagliumi G, Peruga JZ, Brodie BR, Dudek D, Kornowski R, Hartmann F, Gersh BJ, Pocock SJ, Dangas G, Wong SC, Kirtane AJ, Parise H, Mehran R; HORIZONS-AMI Trial Investigators. Bivalirudin during primary PCI in acute myocardial infarction. N Engl J Med. 2008 May 22;358(21):2218-30. doi: 10.1056/NEJMoa0708191. PMID 18499566
- [Background] Lincoff AM, Bittl JA, Harrington RA, Feit F, Kleiman NS, Jackman JD, Sarembock IJ, Cohen DJ, Spriggs D, Ebrahimi R, Keren G, Carr J, Cohen EA, Betriu A, Desmet W, Kereiakes DJ, Rutsch W, Wilcox RG, de Feyter PJ, Vahanian A, Topol EJ; REPLACE-2 Investigators. Bivalirudin and provisional glycoprotein IIb/IIIa blockade compared with heparin and planned glycoprotein IIb/IIIa blockade during percutaneous coronary intervention: REPLACE-2 randomized trial. JAMA. 2003 Feb 19;289(7):853-63. doi: 10.1001/jama.289.7.853. PMID 12588269
- [Background] Stone GW, Ware JH, Bertrand ME, Lincoff AM, Moses JW, Ohman EM, White HD, Feit F, Colombo A, McLaurin BT, Cox DA, Manoukian SV, Fahy M, Clayton TC, Mehran R, Pocock SJ; ACUITY Investigators. Antithrombotic strategies in patients with acute coronary syndromes undergoing early invasive management: one-year results from the ACUITY trial. JAMA. 2007 Dec 5;298(21):2497-506. doi: 10.1001/jama.298.21.2497. PMID 18056903
- [Background] Kinnaird TD, Stabile E, Mintz GS, Lee CW, Canos DA, Gevorkian N, Pinnow EE, Kent KM, Pichard AD, Satler LF, Weissman NJ, Lindsay J, Fuchs S. Incidence, predictors, and prognostic implications of bleeding and blood transfusion following percutaneous coronary interventions. Am J Cardiol. 2003 Oct 15;92(8):930-5. doi: 10.1016/s0002-9149(03)00972-x. PMID 14556868
- [Background] Eikelboom JW, Mehta SR, Anand SS, Xie C, Fox KA, Yusuf S. Adverse impact of bleeding on prognosis in patients with acute coronary syndromes. Circulation. 2006 Aug 22;114(8):774-82. doi: 10.1161/CIRCULATIONAHA.106.612812. Epub 2006 Aug 14. PMID 16908769
- [Background] Manoukian SV, Feit F, Mehran R, Voeltz MD, Ebrahimi R, Hamon M, Dangas GD, Lincoff AM, White HD, Moses JW, King SB 3rd, Ohman EM, Stone GW. Impact of major bleeding on 30-day mortality and clinical outcomes in patients with acute coronary syndromes: an analysis from the ACUITY Trial. J Am Coll Cardiol. 2007 Mar 27;49(12):1362-8. doi: 10.1016/j.jacc.2007.02.027. Epub 2007 Mar 9. PMID 17394970
- [Background] Young E, Prins M, Levine MN, Hirsh J. Heparin binding to plasma proteins, an important mechanism for heparin resistance. Thromb Haemost. 1992 Jun 1;67(6):639-43. PMID 1509402
- [Background] Sobel M, Fish WR, Toma N, Luo S, Bird K, Mori K, Kusumoto S, Blystone SD, Suda Y. Heparin modulates integrin function in human platelets. J Vasc Surg. 2001 Mar;33(3):587-94. doi: 10.1067/mva.2001.112696. PMID 11241131
- [Background] Nikolsky E, Mehran R, Dangas G, Fahy M, Na Y, Pocock SJ, Lincoff AM, Stone GW. Development and validation of a prognostic risk score for major bleeding in patients undergoing percutaneous coronary intervention via the femoral approach. Eur Heart J. 2007 Aug;28(16):1936-45. doi: 10.1093/eurheartj/ehm194. Epub 2007 Jun 15. PMID 17575270
- [Derived] Briguori C, Visconti G, Focaccio A, Donahue M, Golia B, Selvetella L, Ricciardelli B. Novel approaches for preventing or limiting events (Naples) III trial: randomized comparison of bivalirudin versus unfractionated heparin in patients at increased risk of bleeding undergoing transfemoral elective coronary stenting. JACC Cardiovasc Interv. 2015 Mar;8(3):414-423. doi: 10.1016/j.jcin.2014.10.015. Epub 2015 Feb 18. PMID 25703878
- [Derived] Briguori C, Visconti G, Focaccio A, Donahue M, Golia B, Selvetella L, Ricciarelli B. Novel Approaches for Preventing or Limiting Events (NAPLES III) Trial: randomised comparison of bivalirudin versus unfractionated heparin in patients at high risk of bleeding undergoing elective coronary stenting throught the femoral approach. rationale and design. Cardiovasc Drugs Ther. 2014 Jun;28(3):273-9. doi: 10.1007/s10557-014-6518-9. PMID 24781074